CLINICAL TRIAL: NCT01582594
Title: A Registration Study to Evaluate the Performance of CHIRON® RIBA® HCV 3.0 SIA in HCV Antibody Detection
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: OCD-200902
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis C
Keywords: 1000 residual serum/plasma samples; anti-HCV seronegative or seropositive
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A minimum of 1000 qualified specimens shall be collected, including at least 350 anti-HCV seropositive specimens.
  To further evaluate RIBA test specificity in HAV IgG positive, HBsAg positive, HEV IgG positive and anti-HIV positive specimens, approximately 30 specimens of each viral infection will be included in the study.
  A minimum of 60 matched plasma and serum specimens will be collected to evaluate the applicability of the investigational product on different types of samples, including at least 30% of anti-HCV seropositive specimens.
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the accuracy of the CHIRON® RIBA® HCV 3.0 (RIBA, Investigational Product) test using known anti-HCV seropositive and seronegative specimens.

Registration for license application

DETAILED DESCRIPTION:
To evaluate the accuracy of the CHIRON® RIBA® HCV 3.0 (RIBA, Investigational Product) test using known anti-HCV seropositive and seronegative specimens.

To evaluate the effect and applicability of different sample types on RIBA test results through the tests of the investigational product on serum and plasma collected from the same donors.

The specimens with HAV IgG positive, or HBsAg positive, or HEV IgG positive, or anti-HIV positive will be collected and tested for potential interference in the investigational product when used for testing the specimens infected by viruses other than HCV.

This clinical trial is for registration purpose, the study data will be submitted to Regulatory Authority (SFDA) for license application for CHIRON®RIBA®HCV 3.0 SIA reagent.

ELIGIBILITY:
Inclusion Criteria:

* Residual serum or plasma specimens after routine clinical testing; fresh specimens or frozen specimens stored at -20°C or lower within 2 years after collection, with sufficient volume (≥0.5 mL) to complete all the study tests ; 2) Residual serum or plasma specimen is acceptable; matched serum and plasma with EDTA, heparin or citrate used as the anticoagulant. The collection and preparation of the specimens should comply with the standard laboratory operation procedures and the instruction for use (IFU).

Exclusion Criteria:

* Severely hemolytic or turbid specimens; 2) Bacterial contaminated specimens; 3) Specimens that are improperly collected, prepared, or stored or not in accordance with package insert instructions.

Elimination criteria:

1. Errors arising during testing in which the specimen cannot be repeated shall be excluded;
2. Test results that do not pass routine quality control will not be used
3. Any specimen in which the case report form has incomplete data, or the case report form is missing the principal investigator's signature will not be used in the study. Case report forms with missing data will have an explanation for the missing data and should be signed by the principal investigator.
4. Use of unqualified reagents for specimen testing.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The specimens used for this study will be pre-tested by licensed anti-HCV screening methods and / or Nucleic acid test (NAT) in combination with the past history and will be classified as either seronegative or seropositive.
Sampling Method: Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of the CHIRON® RIBA® HCV 3.0 | up to 30 weeks
  To evaluate the accuracy of the CHIRON® RIBA® HCV 3.0 (RIBA, Investigational Product) test using known anti-HCV seropositive and seronegative specimens. As the study early terminated,no evaluation performed.

SECONDARY OUTCOMES:
the effect and applicability of different sample types on RIBA test results | up to 30 weeks
  To evaluate the effect and applicability of different sample types on RIBA test results through the tests of the investigational product on serum and plasma collected from the same donors.As the study early terminated,no evaluation performed.
potential interference in RIBA | up to 30 weeks
  The specimens with HAV IgG positive, or HBsAg positive, or HEV IgG positive, or anti-HIV positive will be collected and tested for potential interference in the investigational product when used for testing the specimens infected by viruses other than HCV. As the study early terminated,no evaluation performed.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanli Mao, Professor, Principal Investigator — Beijing 302 Hospital; Yanping Luo, Professor, Principal Investigator — Chinese PLA General Hospital; Xinxin Zhang, Professor, Principal Investigator — Ruijin Hospital; Tai Guo, Director, Principal Investigator — National Institites of Food and Drug control
Locations (4):
- China (4):
  - 302 military hospital of China, Beijing, Beijing Municipality
  - National institues for Food and Drug control, Beijing, Beijing Municipality
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - Ruijin hospital Shanghai Jiaotong University school of medicine, Shanghai